CLINICAL TRIAL: NCT02051998
Title: Analysis of the Directional Spread of Geographic Atrophy (GA) in Patients With Age-related Macular Degeneration (AMD)
Brief Title: Directional Spread in Geographic Atrophy
Acronym: DSGA
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Prof. Dr. Monika Fleckenstein, MD, Prof. Dr. med., University Hospital, Bonn
Other Study IDs: FL 658/4-1 and FL 658/4-2
Record Dates: First submitted 2014-01-08; First posted 2014-01-31 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Nonexudative Age-related Macular Degeneration
Keywords: Geographic atrophy; Age-related macular degeneration; Retina; Retinal pigment epithelium; Optical coherence tomography; Scanning laser ophthalmoscopy
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of irreversible blindness in industrial countries. In the late stages of the disease, neovascular changes or the development of geographic atrophy (GA) may induce severe visual loss. GA is characterized by the development of areas of outer retinal atrophy with continuous spread over time that is corresponded to an visual field defect for the patient. The pathogenesis is still incompletely understood. Despite the break-through in the treatment of neovascular AMD by intravitreally administrated vascular endothelial growths factor (VEGF) inhibitors, there is yet no treatment available to slow down or halt the disease process in GA. We and others have demonstrated that the total GA area progression shows large differences between patients. Potential factors influencing differential progression have been intensely studied: While neither systemic nor genetic factors have been shown to influence GA progression, ocular characteristics such as GA baseline size or phenotypic features of fundus autofluorescence (FAF) abnormalities have been identified as risk characteristics for increased GA progression. While these previous studies have mainly focused on the characterization of total GA area progression, topographic directional spread has not been analyzed and relevant predictive markers are yet unknown. There may be large differences in the local GA progression. The primary objective of this study is to identify specific characteristics, for the local GA progression. The knowledge of such risk factors may help to better understand the pathogenesis of GA. The identification of predictive markers will allow for better prognostic assessment of the individual disease process. The DSGA study is the extension trial of the FAM (Fundus Autofluorescence in Age-related Macular Degeneration) study (NCT00393692).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Men and women, any race, aged 55 years or older at the baseline visit
* If both eyes meet the criteria to be study eye either eye will be included into the analysis.
* Patient is willing to undergo ocular examinations once every 6 for up to 24 months

Exclusion Criteria:

* The presence or history of CNV (choroidal neovascular membrane) in the study eye
* Ocular disease in the study eye that may confound assessment of the retina, other than non-exudative AMD (e.g., diabetic retinopathy, uveitis)
* Any systemic disease with a limited survival prognosis (e.g., cancer, severe/unstable cardiovascular disease).
* Any condition that would make adherence to the examination schedule of once every 6 months for up to 24 months difficult or unlikely, e.g., personality disorder, chronic alcoholism, Alzheimer's Disease or drug abuse
* Known medical history of allergy or sensitivity to tropicamide or fluorescein dye that is clinically relevant in the investigator's opinion

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable for the study will be recruited at the University of Bonn, Department of Ophthalmology
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2013-06; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Change of geographic atrophy size to baseline | 24 months

SECONDARY OUTCOMES:
Change in BCVA from baseline | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fleckenstein, Prof. Dr. med., Principal Investigator — Department of Ophthalmology, University of Bonn
Locations (1):
- Department of Ophthalmology, University of Bonn, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Holz FG, Bindewald-Wittich A, Fleckenstein M, Dreyhaupt J, Scholl HP, Schmitz-Valckenberg S; FAM-Study Group. Progression of geographic atrophy and impact of fundus autofluorescence patterns in age-related macular degeneration. Am J Ophthalmol. 2007 Mar;143(3):463-72. doi: 10.1016/j.ajo.2006.11.041. Epub 2006 Dec 22. PMID 17239336
- [Background] Schmitz-Valckenberg S, Bultmann S, Dreyhaupt J, Bindewald A, Holz FG, Rohrschneider K. Fundus autofluorescence and fundus perimetry in the junctional zone of geographic atrophy in patients with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4470-6. doi: 10.1167/iovs.03-1311. PMID 15557456
- [Background] Fleckenstein M, Adrion C, Schmitz-Valckenberg S, Gobel AP, Bindewald-Wittich A, Scholl HP, Mansmann U, Holz FG; FAM Study Group. Concordance of disease progression in bilateral geographic atrophy due to AMD. Invest Ophthalmol Vis Sci. 2010 Feb;51(2):637-42. doi: 10.1167/iovs.09-3547. Epub 2009 Sep 24. PMID 19797219
- [Background] Schmitz-Valckenberg S, Brinkmann CK, Alten F, Herrmann P, Stratmann NK, Gobel AP, Fleckenstein M, Diller M, Jaffe GJ, Holz FG. Semiautomated image processing method for identification and quantification of geographic atrophy in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2011 Sep 29;52(10):7640-6. doi: 10.1167/iovs.11-7457. PMID 21873669
- [Background] Fleckenstein M, Charbel Issa P, Helb HM, Schmitz-Valckenberg S, Finger RP, Scholl HP, Loeffler KU, Holz FG. High-resolution spectral domain-OCT imaging in geographic atrophy associated with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2008 Sep;49(9):4137-44. doi: 10.1167/iovs.08-1967. Epub 2008 May 16. PMID 18487363
- [Background] Fleckenstein M, Schmitz-Valckenberg S, Adrion C, Kramer I, Eter N, Helb HM, Brinkmann CK, Charbel Issa P, Mansmann U, Holz FG. Tracking progression with spectral-domain optical coherence tomography in geographic atrophy caused by age-related macular degeneration. Invest Ophthalmol Vis Sci. 2010 Aug;51(8):3846-52. doi: 10.1167/iovs.09-4533. Epub 2010 Mar 31. PMID 20357194
- [Background] Fleckenstein M, Schmitz-Valckenberg S, Martens C, Kosanetzky S, Brinkmann CK, Hageman GS, Holz FG. Fundus autofluorescence and spectral-domain optical coherence tomography characteristics in a rapidly progressing form of geographic atrophy. Invest Ophthalmol Vis Sci. 2011 Jun 1;52(6):3761-6. doi: 10.1167/iovs.10-7021. PMID 21310912
- [Background] Schmitz-Valckenberg S, Fleckenstein M, Helb HM, Charbel Issa P, Scholl HP, Holz FG. In vivo imaging of foveal sparing in geographic atrophy secondary to age-related macular degeneration. Invest Ophthalmol Vis Sci. 2009 Aug;50(8):3915-21. doi: 10.1167/iovs.08-2484. Epub 2009 Apr 1. PMID 19339734
- [Derived] Kunzel SH, Broadbent E, Moller PT, Lindner M, Goerdt L, Czauderna J, Schmitz-Valckenberg S, Holz FG, Pfau M, Fleckenstein M. Association of Lesion Location and Functional Parameters with Vision-Related Quality of Life in Geographic Atrophy Secondary to Age-related Macular Degeneration. Ophthalmol Retina. 2024 Aug;8(8):794-803. doi: 10.1016/j.oret.2024.01.025. Epub 2024 Feb 3. PMID 38311207
- [Derived] Kunzel SH, Moller PT, Lindner M, Goerdt L, Nadal J, Schmid M, Schmitz-Valckenberg S, Holz FG, Fleckenstein M, Pfau M. Determinants of Quality of Life in Geographic Atrophy Secondary to Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2020 May 11;61(5):63. doi: 10.1167/iovs.61.5.63. PMID 32462198
- [Derived] Pfau M, von der Emde L, Dysli C, Thiele S, Moller PT, Lindner M, Nadal J, Schmid M, Schmitz-Valckenberg S, Holz FG, Fleckenstein M. Light Sensitivity Within Areas of Geographic Atrophy Secondary to Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2019 Sep 3;60(12):3992-4001. doi: 10.1167/iovs.19-27178. PMID 31560765
- [Derived] Pfau M, Lindner M, Goerdt L, Thiele S, Nadal J, Schmid M, Schmitz-Valckenberg S, Sadda SR, Holz FG, Fleckenstein M; Fundus Autofluorescence in Age-Related Macular Degeneration Study Group. PROGNOSTIC VALUE OF SHAPE-DESCRIPTIVE FACTORS FOR THE PROGRESSION OF GEOGRAPHIC ATROPHY SECONDARY TO AGE-RELATED MACULAR DEGENERATION. Retina. 2019 Aug;39(8):1527-1540. doi: 10.1097/IAE.0000000000002206. PMID 29781974
- [Derived] Lindner M, Kosanetzky S, Pfau M, Nadal J, Gordt LA, Schmitz-Valckenberg S, Schmid M, Holz FG, Fleckenstein M; FAM-Study Group. Local Progression Kinetics of Geographic Atrophy in Age-Related Macular Degeneration Are Associated With Atrophy Border Morphology. Invest Ophthalmol Vis Sci. 2018 Mar 20;59(4):AMD12-AMD18. doi: 10.1167/iovs.17-23203. PMID 29558533
- [Derived] Fleckenstein M, Mitchell P, Freund KB, Sadda S, Holz FG, Brittain C, Henry EC, Ferrara D. The Progression of Geographic Atrophy Secondary to Age-Related Macular Degeneration. Ophthalmology. 2018 Mar;125(3):369-390. doi: 10.1016/j.ophtha.2017.08.038. Epub 2017 Oct 27. PMID 29110945
- [Derived] Lindner M, Nadal J, Mauschitz MM, Luning A, Czauderna J, Pfau M, Schmitz-Valckenberg S, Holz FG, Schmid M, Fleckenstein M. Combined Fundus Autofluorescence and Near Infrared Reflectance as Prognostic Biomarkers for Visual Acuity in Foveal-Sparing Geographic Atrophy. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO61-BIO67. doi: 10.1167/iovs.16-21210. PMID 28475704
- [Derived] Lindner M, Bezatis A, Czauderna J, Becker E, Brinkmann CK, Schmitz-Valckenberg S, Fimmers R, Holz FG, Fleckenstein M. Choroidal thickness in geographic atrophy secondary to age-related macular degeneration. Invest Ophthalmol Vis Sci. 2015 Jan 13;56(2):875-82. doi: 10.1167/iovs.14-14933. PMID 25587059
- See also: Webpage of the University Eye Hospital of Bonn — http://www.augenklinik.uni-bonn.de/